CLINICAL TRIAL: NCT03618953
Title: Phase 1/1b, Multicenter, Open-label Trial of Oncolytic MG1 Virus (MG1-E6E7) With Adenovirus Vaccine (Ad-E6E7) Both Expressing Mutant Human Papilloma Virus (HPV) E6 and E7 and Atezolizumab in Pts With HPV Assoc. Cancers
Brief Title: This is a Trial of MG1-E6E7 With Ad-E6E7 and Atezolizumab in Patients With HPV Associated Cancers
Acronym: Kingfisher
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Virus potency titer of drug product as determined by an improved potency assay was lower than originally determined by the assay described in the IND.
Sponsor: Turnstone Biologics, Corp. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Ad-MG1-E6E7-002
Record Dates: First submitted 2018-06-22; First posted 2018-08-07 (Actual); Last update posted 2023-04-14 (Actual); Status verified 2023-04

CONDITIONS: HPV-Associated Cancers
MeSH Terms: interventions — atezolizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm 1 (Intravenous dosing) (Experimental): Fixed dose of Ad-E6E7 administered IM on study Day 1. Followed by one of 3 dose levels (escalation) of MG1-E6E7 administered as 4 infusion (IV) doses over 2 weeks starting at study day 15.
  Fixed dose of atezolizumab administered IV every 3weeks starting at study day 43.
  Interventions: Biological: Ad-E6E7; Biological: MG1-E6E7; Biological: Atezolizumab
- Arm 2 (Intravenous and Intra-tumoral injection dosing) (Experimental): Fixed dose of Ad-E6E7 administered IM on study Day 1. Followed by one of 2 dose levels (escalation) of MG1-E6E7 administered as 1 IV dose, starting at study day 15, followed by 2 intratumoral (IT) doses administered on study days 18 & 29.
  Fixed dose of atezolizumab administered IV every 3weeks starting at study day 43.
  Interventions: Biological: Ad-E6E7; Biological: MG1-E6E7; Biological: Atezolizumab

INTERVENTIONS:
Biological: Ad-E6E7 — Adenovirus vaccine expressing mutant HPV E6 and E7
Biological: MG1-E6E7 — MG1 Maraba oncolytic virus expressing mutant HPV E6 and E7
Biological: Atezolizumab — monoclonal antibody; checkpoint inhibitor
  Other Names: Tecentriq

SUMMARY:
This is a Phase 1/1b open-label dose escalation trial of Ad/MG1-E6E7 and sequential treatment with atezolizumab in patients with HPV associated cancers. This study will consist of two arms. Both arms will dose escalate (MG1-E6E7) using a 3 + 3 design in Phase 1 to establish initial safety and the maximum tolerated dose (MTD) / maximum feasible dose (MFD).

* Arm 1 - intravenous (IV) administration of MG1-E6E7 following intramuscular (IM) AD-E6E7 priming and subsequent treatment with IV atezolizumab.
* Arm 2 - intratumoral (IT) and IV injection of MG1-E6E7 following (IM) Ad-E6E7 priming and subsequent treatment with IV atezolizumab.

In the Phase 1b expansion for each arm, additional patients will be enrolled at the MTD as determined in Phase 1 in order to more thoroughly explore immune response, pharmacokinetics/dynamics, and safety for the patient populations with Cervical cancer, HPV positive (HPV+) Oropharyngeal cancer (Phase 1B, Arm 1, Cohorts A and B respectively) and HPV+ tumors with injectable lesions (Phase 1B, Arm 2, Cohort 3).

ELIGIBILITY:
Key Inclusion Criteria:

* Histologically or cytologically confirmed recurrent or metastatic HPV associated tumor (cervical, oropharyngeal, vulvar, vaginal, anal, or penile) with documented disease progression.
* Arm 1, Phase 1 dose escalation: Cervical, HPV+ oropharyngeal, vulvar, vaginal, anal, or penile
* Arm 1, Cohort A: Cervical cancer
* Arm 1, Cohort B: HPV+ Oropharyngeal cancer
* Arm 2 Phase 1 dose escalation and Cohort C: Cervical, oropharyngeal, vulvar, vaginal, anal, or penile
* Failed, refused or intolerant to systemic therapy
* Measurable disease based on RECIST 1.1
* At least one tumor mass amenable to core needle biopsy
* Arm 2 only: At least one tumor judged as being safely injectable
* ECOG performance status 0 or 1
* Demonstrate adequate organ function
* Additional Inclusion criteria exist

Key Exclusion Criteria:

* Prior systemic therapy within 4 weeks.
* Patients receiving prior XRT must have recovered from any acute toxicity.
* Currently receiving/received experimental therapy within 4 weeks.
* Prior treatment with any HPV vaccine therapy for cancer.
* Requires use of anti-platelet or anti-coagulant therapy that cannot be safely suspended for per protocol biopsies or intra-tumoral injections.
* Known active CNS metastases and/or carcinomatous meningitis.
* Clinically significant tumor invasion/ rapidly accumulating ascites, pericardial or pleural effusions.
* Active infection requiring systemic therapy.
* Active autoimmune disease that has required systemic therapy in the past 2 years.
* Conditions likely to have resulted in splenic dysfunction.
* Known HIV/AIDS, active HBV or HCV infection.
* Received prior treatment with vesicular stomatitis (VSV) viral vector.
* Received immunosuppressive medication within 4 weeks. (>10mg/day prednisone)
* ≥ Grade 2 dyspnea and/or require supplemental oxygen
* Known intolerance to anti-PD-1 or anti-PD-L1 antibody therapy
* Additional Exclusion criteria exist

Exclusion Criteria Household Contacts:

* Patients with household contacts meeting any of the following criteria are ineligible for study entry unless alternate living arrangements can be made, while under contact precautions.
* Women who are pregnant or nursing an infant
* Children < 1 year old
* Individuals who are severely immunocompromised
* Contact precautions are from initial treatment with MG1-E6E7 to 7 days after the last dose of MG1-E6E7

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2018-06-21 (Actual); Primary Completion 2021-03-05 (Actual); Study Completion 2021-03-05 (Actual)

PRIMARY OUTCOMES:
Safety of Ad/MG1-E6E7 administration in HPV associated cancers | 8 months
  Safety will be determined by assessing the severity and frequency of treatment emergent Adverse Events and clinical laboratory toxicity using NCI CTCAE v 4.03.
Determine the maximum tolerated dose (MTD)/ maximum feasible dose (MFD) of Ad/MG1-E6E7 in HPV associated cancers | 4 to 6 weeks after first treatment with Ad/MG1-E6E7
  MTD/MFD of Ad/MG1-E6E7 administered by IV infusion alone and IV infusion followed by direct injection of tumor (IT injection) in HPV associated cancers

SECONDARY OUTCOMES:
Concentration of Ad/MG1-E6E7 in blood | 4 to 6 weeks after first treatment with Ad/MG1-E6E7
  Change over time in the number of MG1-E6E7 genomes (qPCR) and MG1-E6E7 infectious units (PFU) in blood
Assess for the biodistribution and shedding of Ad/MG1-E6E7 | 6 weeks after first treatment with Ad/MG1-E6E7
  Determine if there is any shedding of Ad/MG1-E6E7 into the environment by detecting the presence of viral plaque forming units (PFUs) in urine samples, cheek swabs, and rectal swabs after Ad/MG1-E6E7 treatment
Measure the differences in pre- and post treatment levels of T cell subsets and T cell activation status | Before and after each dose of Ad/MG1-E6E7 and then every 3 weeks until treatment discontinuation
  Analyze the change over time in the the frequencies, absolute numbers and subsets of T cells (including regulatory T cells)
Anti-tumor activity | Every 6 weeks for the first course of treatment and then every 9 weeks until date of documented progression by irRECIST, up to 2 years
  Evaluate tumor response by CT scan using RECIST v1.1 and irRECIST criteria in the overall patient population and the HPV16/18 positive patient population

CONTACTS AND LOCATIONS:
Overall Officials: Steve Bernstein, MD, Study Director — Turnstone Biologics
Locations (8):
- United States (5):
  - University of Miami, Miami, Florida
  - Billings Clinic, Billings, Montana
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - University of Toledo-The Eleanor N. Dana Cancer Center, Toledo, Ohio
  - University of Texas-MD Anderson Cancer Center, Houston, Texas
- Canada (3):
  - Juravinski Cancer Centre, Hamilton, Ontario
  - Ottawa Hospital Research Institute, Ottawa, Ontario
  - Princess Margaret Hospital, Toronto, Ontario